CLINICAL TRIAL: NCT02006680
Title: Markers of Adequate Pubertal Suppression During Supprelin LA Therapy for Central Precocious Puberty
Brief Title: Markers of Pubertal Suppression During Therapy for Precocious Puberty
Status: Terminated | Type: Observational
Why Stopped: Inadequate Recruitment
Sponsor: University of Minnesota (Other)
Collaborators: Endo Pharmaceuticals (Industry); Atlantic Center for Research (Unknown); Goryeb Children's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1303M29681
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Central Precocious Puberty
Keywords: Central Precocious Puberty; Suppression; Alpha Subunit; Leuprolide Stimulation Test
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum will be collected at four different time points.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children with Central Precocious Puberty: Children with Central Precocious Puberty will have hormonal testing of markers of puberty up to 30 days prior to placement of a Supprelin LA insert and 28-97 days after placement of the Supprelin LA insert.

SUMMARY:
The best way to measure whether treatment of children with central precocious puberty is working is to do a hormone stimulation test (leuprolide stimulation test) that requires injection of a medication and multiple blood draws to see if the hormonal response is suppressed (blocked). The hypothesis of this study is that random measurement of the free alpha subunit of pituitary glycoprotein, a protein related to the pituitary hormones that stimulate puberty, will provide an adequate alternative to the leuprolide stimulation testfor monitoring efficacy of pubertal suppression with Supprelin LA®.

DETAILED DESCRIPTION:
During clinical trials of Supprelin LA®, leuprolide stimulation tests were performed to determine adequacy of suppression. However, the use of this stimulation test to monitor suppression requires an expensive medication and collection of multiple blood samples. Alternative methods of monitoring pubertal suppression during gonadotropin releasing hormone receptor agonist (GnRHa) therapy have included both random and trough levels of Luteinizing Hormone (LH), estradiol or inhibin B. Recently, the free alpha subunit of pituitary glycoprotein (FASPG) has also been shown to be a potentially useful marker of hormonal suppression (Hirsch HJ, et al, JCEM 95:2841, 2010) as it undergoes a paradoxical rise following initiation of therapy, and reverts to baseline upon completion.

In this investigator-initiated pilot study we will evaluate novel markers of pubertal suppression in children receiving standard of care gonadotropin releasing hormone receptor agonist therapy for the treatment of central precocious puberty. Children with central precocious puberty who have selected treatment with Supprelin LA will undergo hormonal testing of markers of pubertal activity before and after placement of the Supprelin LA insert.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age: 3 to 9 years old, inclusive
* Diagnosis of Central Precocious or Rapidly Progressive Puberty
* Bone Age more than 1 year advanced (obtained within 6 months of screening) AND
* Breasts Tanner II or greater AND
* One of the following:
* Random LH > 1 mIU/mL
* Leuprolide-stimulated LH > 4 mIU/mL
* Random estradiol > 20 pg/mL
* Leuprolide-stimulated 24 hour estradiol >20 pg/mL
* Naïve to GnRHa therapy
* Approved to receive Supprelin LA® therapy
* Have an acceptable surrogate capable of giving consent on the subject's behalf.

Exclusion Criteria:

* Previous GnRHa therapy
* Presence of peripheral precocious puberty including CAH

Ages: 3 Years to 9 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Females diagnosed with central precocious puberty or rapidly progressive puberty based upon age at start of puberty, physical examination, serum hormone levels and bone age X-Ray will be recruited. This will be a convenience sample of children scheduled to receive Supprelin LA insert placement. The subjects will be recruited from two pediatric endocrinology clinic systems.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of free alpha subunit of pituitary glycoprotein to identify subjects with appropriate pubertal suppression. | Up to 12 months
  The primary outcome of the study will be the sensitivity and specificity of a subject having elevated random FASPG values (> 0.6 ng/mL) to identify subjects who are appropriately suppressed based upon a leuprolide-stimulated LH <4 mIU/mL. This outcome will be based upon results of puberty hormone suppression testing obtained 28-97 days after placement of the Supprelin LA insert.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Miller, MD, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Atlantic Center for Research, Morristown, New Jersey